CLINICAL TRIAL: NCT03534141
Title: Mild Hypothermia and Acute Kidney Injury in Liver Transplantation (MHALT) Trial
Brief Title: Mild Hypothermia and Acute Kidney Injury in Liver Transplantation
Acronym: MHALT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated 9/24/23 at 85% target enrollment due to slow accrual of subjects. The decline in enrollment was attributed to changing surgical demographics (higher MELD, more DCD grafts, and increasing use of Normothermic Perfusion technology).
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Colorado, Denver (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-22384
Record Dates: First submitted 2018-04-27; First posted 2018-05-23 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis; End Stage Liver Disease; Acute Kidney Injury; Liver Transplant; Complications; Chronic Kidney Diseases; Hepatitis c; Hepatitis B; NASH - Nonalcoholic Steatohepatitis; Alcoholic Cirrhosis; Hepatocellular Carcinoma
Keywords: Hypothermia; NGAL - Neutrophil Gelatinase-associated Lipocalin
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease; Acute Kidney Injury; Renal Insufficiency, Chronic; Hepatitis C; Hepatitis B; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis, Alcoholic; Carcinoma, Hepatocellular; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mild hypothermia & Esophageal cooling/warming device (Experimental): The target core temperature is 34-35 °C.
  Interventions: Device: Esophageal cooling/warming device; Other: Mild hypothermia
- Normothermia & Esophageal cooling/warming device (Active Comparator): The target core temperature is 36.5-37.5 °C.
  Interventions: Device: Esophageal cooling/warming device; Other: Normothermia

INTERVENTIONS:
Device: Esophageal cooling/warming device — The EnsoETM (formerly known as Esophageal Cooling Device) is a non-sterile multilumen silicone tube placed in the esophagus for the purpose of cooling or warming a patient while allowing gastric decompression and drainage. It is placed in a manner identical to a standard orogastric tube, which is standard equipment for liver transplant surgery. It is removed at the end of surgery. Control of the patient's temperature is achieved by connecting the EnsoETM to an external heat exchanger (Gaymar Medi-Therm III or similar system). The Medi-Therm III is a standard device used in operating rooms for warming patients with a conductive table warming pad. The Medi-Therm III circulates temperature-controlled water through a closed-loop system via the two outer lumens of the EnsoETM. Water temperature ranges from 4°C - 42°C.
  Other Names: EnsoETM; ECD - Esophageal Cooling Device
Other: Mild hypothermia — Cooling will be initiated after induction of anesthesia and maintained throughout the anhepatic phase of liver transplantation. In all feasible cases the surgeon will cover the peritoneal surface over the right kidney, which is exposed during the operation, with ice-cold sponges to enhance cooling of the renal parenchyma. After blood flow is completely restored to the liver, the esophageal cooling device and other standard measures (forced-air, fluid, and table warmers, plus a heated anesthesia circuit) will be used to actively re-warm the patient (expected warming rate ≥ 1 deg C/hour). The goal is to achieve normothermia by case end.
  Arms: Mild hypothermia & Esophageal cooling/warming device
Other: Normothermia — After induction of anesthesia, the esophageal cooling/warming device and standard warming measures will be used to maintain normothermia throughout the operation.
  Arms: Normothermia & Esophageal cooling/warming device

SUMMARY:
Acute kidney injury (AKI), or worsening kidney function, is a common complication after liver transplantation (20-90% in published studies). Patients who experience AKI after liver transplantation have higher mortality, increased graft loss, longer hospital and intensive care unit stays, and more progression to chronic kidney disease compared with those who do not. In this study, half of the participants will have their body temperature cooled to slightly lower than normal (mild hypothermia) for a portion of the liver transplant operation, while the other half will have their body temperature maintained at normal. The study will evaluate if mild hypothermia protects from AKI during liver transplantation.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of mild hypothermia during liver transplantation to provide protection from AKI. Participants will be randomized to normothermia (36.5-37.5 °C) versus mild hypothermia (34-35 °C) during a portion of the liver transplant operation. The protocol is based on preliminary data from rodent models showing that hypothermia protects the kidneys from ischemia-reperfusion injury, as well as studies in deceased organ donors showing that cooling improves post-transplant organ function. Temperature will be maintained with standard techniques plus a minimally-invasive esophageal cooling device that is approved by the U.S. Food and Drug Administration. The investigators hypothesize that mild hypothermia will reduce the incidence and severity of AKI after liver transplantation(LTx). Standard surrogates (e.g., change in serum creatinine, need for initiation of dialysis) and biomarkers will be used to assess the severity of kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation from a donor after neurologic determination of death

Exclusion Criteria:

* Liver transplantation from a donor after cardiac death
* Acute liver failure
* Living-donor liver transplantation
* Simultaneous liver-kidney transplantation
* Preoperative renal replacement therapy
* Preoperative intubation
* Portopulmonary hypertension
* Machine perfusion of liver graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Bokoch, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niemann CU, Feiner J, Swain S, Bunting S, Friedman M, Crutchfield M, Broglio K, Hirose R, Roberts JP, Malinoski D. Therapeutic Hypothermia in Deceased Organ Donors and Kidney-Graft Function. N Engl J Med. 2015 Jul 30;373(5):405-14. doi: 10.1056/NEJMoa1501969. PMID 26222557
- [Background] Angeli P, Gines P, Wong F, Bernardi M, Boyer TD, Gerbes A, Moreau R, Jalan R, Sarin SK, Piano S, Moore K, Lee SS, Durand F, Salerno F, Caraceni P, Kim WR, Arroyo V, Garcia-Tsao G; International Club of Ascites. Diagnosis and management of acute kidney injury in patients with cirrhosis: revised consensus recommendations of the International Club of Ascites. Gut. 2015 Apr;64(4):531-7. doi: 10.1136/gutjnl-2014-308874. Epub 2015 Jan 28. No abstract available. PMID 25631669
- [Background] Niemann CU, Walia A, Waldman J, Davio M, Roberts JP, Hirose R, Feiner J. Acute kidney injury during liver transplantation as determined by neutrophil gelatinase-associated lipocalin. Liver Transpl. 2009 Dec;15(12):1852-60. doi: 10.1002/lt.21938. PMID 19938135
- [Background] Kalasbail P, Makarova N, Garrett F, Sessler DI. Heating and Cooling Rates With an Esophageal Heat Exchange System. Anesth Analg. 2018 Apr;126(4):1190-1195. doi: 10.1213/ANE.0000000000002691. PMID 29283916
- [Background] Karapanagiotou A, Dimitriadis C, Papadopoulos S, Kydona C, Kefsenidis S, Papanikolaou V, Gritsi-Gerogianni N. Comparison of RIFLE and AKIN criteria in the evaluation of the frequency of acute kidney injury in post-liver transplantation patients. Transplant Proc. 2014 Nov;46(9):3222-7. doi: 10.1016/j.transproceed.2014.09.161. PMID 25420865
- [Background] Kellum JA, Zarbock A, Nadim MK. What endpoints should be used for clinical studies in acute kidney injury? Intensive Care Med. 2017 Jun;43(6):901-903. doi: 10.1007/s00134-017-4732-1. Epub 2017 Mar 2. No abstract available. PMID 28255614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between July 2018 and August 2023 from patients scheduled for deceased donor liver transplantation at three transplant centers.
Pre-assignment Details: Participants were enrolled after liver transplantation was scheduled but before entering the operating room for surgery. Before proceeding with randomization, it was necessary for the attending surgeon to verify that the liver graft was suitable for transplantation. If that was not the case, the transplant could be aborted before randomization.
Groups:
- Mild Hypothermia & Esophageal Cooling/Warming Device: The target core temperature is 34-35 °C.
  Esophageal cooling/warming device: The EnsoETM (formerly known as Esophageal Cooling Device) is a non-sterile multilumen silicone tube placed in the esophagus for the purpose of cooling or warming a patient while allowing gastric decompression and drainage. It is placed in a manner identical to a standard orogastric tube and is removed at the end of surgery. Control of the patient's temperature is achieved by connecting the EnsoETM to an external heat exchanger (Gaymar Medi-Therm III or similar system). The Medi-Therm III circulates temperature-controlled water through a closed-loop system via the two outer lumens of the EnsoETM. Water temperature ranges from 4°C - 42°C.
  Mild hypothermia: Cooling will be initiated after induction of anesthesia and maintained throughout the anhepatic phase of liver transplantation. In all feasible cases the surgeon will cover the peritoneal surface over the right kidney, which is exposed during the operation, with ice-cold sponges to enhance cooling of the renal parenchyma. After blood flow is completely restored to the liver, the esophageal cooling device and other standard measures (forced-air, fluid, and table warmers, plus a heated anesthesia circuit) will be used to actively re-warm the patient (expected warming rate ≥ 1 deg C/hour). The goal is to achieve normothermia by case end.
Period: Overall Study
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Started | 87 | 88
Completed | 86 | 85
Not Completed | 1 | 3
Not completed — Enrolled in other clinical trial | 1 | 0
Not completed — Liver transplant aborted after randomization | 0 | 2
Not completed — Liver graft explanted due to surgical issue | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 64] | 59 [52 to 65] | 59 [51 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 51 | 58 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 28 | 54
  Not Hispanic or Latino | 60 | 57 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 3 | 1 | 4
  White | 57 | 55 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 19 | 34
Region of Enrollment [Number; unit: participants]
  United States | 86 | 85 | 171
Etiology of liver disease [Count of Participants; unit: Participants]
  Hepatitis C | 17 | 13 | 30
  Hepatitis B | 6 | 3 | 9
  Alcoholic | 22 | 30 | 52
  Nonalcoholic steatohepatitis (NASH) | 20 | 21 | 41
  Cryptogenic | 2 | 8 | 10
  Other | 19 | 10 | 29
Model for End-stage Liver Disease-Sodium score [Median (Inter-Quartile Range); unit: units on a scale] — This score reflects the severity of liver disease and is used to determine priority for liver transplantation. It is a standard assessment for patients with liver disease calculated from the preoperative serum sodium, total bilirubin, international normalized ratio, and creatinine (or the need for preoperative renal replacement therapy). The scale ranges from 6-40, with higher scores representing more severe liver disease. For additional details and full calculation, please see Kim WR et al. N Engl J Med 2008;359:1018-1026.
  units on a scale | 21 [14 to 29] | 22 [14 to 28] | 22 [14 to 28]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.6 [24.7 to 31.1] | 27.2 [23.7 to 30.2] | 27.3 [24.0 to 31.0]

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury (AKI)
Description: Acute Kidney Injury (AKI) is defined according to the International Club for Ascites (ICA) 2015 criteria, a revision of the Kidney Disease Improving Global Outcome (KDIGO) criteria for patients with cirrhosis (Angeli P, Ginès P, Wong F, Bernardi M, Boyer TD, Gerbes A, et al. Gut. 2015 Apr;64(4):531-7). AKI is defined as an increase in sCr ≥ 0.3 mg/dL within 48 hours, or a percentage increase ≥ 50% from baseline, or the initiation of renal replacement therapy. Baseline creatinine is defined as the most recent value obtained prior to liver transplantation.
Time Frame: 72 hours from the end of surgery
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Mild Hypothermia & Esophageal Cooling/Warming Device: The target core temperature is 34-35 °C.
  Esophageal cooling/warming device: The EnsoETM (formerly known as Esophageal Cooling Device) is a non-sterile multilumen silicone tube placed in the esophagus for the purpose of cooling or warming a patient while allowing gastric decompression and drainage. It is placed in a manner identical to a standard orogastric tube. It is removed at the end of surgery. Control of the patient's temperature is achieved by connecting the EnsoETM to an external heat exchanger (Gaymar Medi-Therm III or similar system). The Medi-Therm III circulates temperature-controlled water through a closed-loop system via the two outer lumens of the EnsoETM. Water temperature ranges from 4°C - 42°C.
  Mild hypothermia: Cooling will be initiated after induction of anesthesia and maintained throughout the anhepatic phase of liver transplantation. In all feasible cases the surgeon will cover the peritoneal surface over the right kidney, which is exposed during the operation, with ice-cold sponges to enhance cooling of the renal parenchyma. After blood flow is completely restored to the liver, the esophageal cooling device and other standard measures (forced-air, fluid, and table warmers, plus a heated anesthesia circuit) will be used to actively re-warm the patient (expected warming rate ≥ 1 deg C/hour). The goal is to achieve normothermia by case end.
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
Participants | 56 | 47

2. Secondary Outcome: Distribution of the Stages of Acute Kidney Injury (AKI)
Description: The International Club for Ascites (ICA) 2015 criteria, a revision of the Kidney Disease Improving Global Outcome (KDIGO) criteria for patients with cirrhosis (Angeli P, Ginès P, Wong F, Bernardi M, Boyer TD, Gerbes A, et al. Gut. 2015 Apr;64(4):531-7), will be used to define the stage of AKI (Stage 1, 2, or 3). The distribution of the stages of AKI within 72 hours after liver transplantation. The stages of AKI are defined as follows based on the serum creatinine (sCr):
  AKI Stage 1: increase in sCr ≥ 0.3 mg/dL, or an increase in sCr ≥ 1.5-fold and ≤ 2-fold from baseline.
  AKI Stage 2: increase in sCr > 2-fold and ≤ 3-fold from baseline. AKI Stage 3: increase in sCr > 3-fold from baseline, or sCr ≥ 4.0 with an acute increase of ≥ 0.3 mg/dL, or initiation of renal replacement therapy.
Time Frame: 72 hours from the end of surgery
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
Participants
  No AKI | 30 | 38
  AKI Stage 1 | 32 | 20
  AKI Stage 2 | 13 | 9
  AKI Stage 3 | 11 | 18

3. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: Time after liver transplantation until patient is discharged from the ICU to a regular hospital bed.
Time Frame: Time from end of liver transplant to ICU discharge, approximately 1 to 3 days
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
hours | 36 [0 to 70] | 37 [19 to 68]

4. Secondary Outcome: Duration of Hospital Stay
Description: From the date of liver transplantation until the date patient is discharged from the hospital.
Time Frame: Time from liver transplant to hospital discharge, approximately 1-2 weeks.
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
days | 7 [5 to 9] | 7 [5 to 10]

5. Secondary Outcome: Patient Survival
Description: From the date of liver transplantation until the date of death from any cause.
Time Frame: up to 1 year
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
Participants | 81 | 78

6. Secondary Outcome: Need for Renal Replacement Therapy
Description: Patient is receiving continuous renal replacement therapy or dialysis at the time of follow-up. If patient died before the indicated follow-up time, the outcome was counted as positive (patient was on renal replacement therapy).
Time Frame: 72 hours, 30 days, and 1 year. The original protocol specified assessment at 1 week after surgery. However, this data was unable to be collected and we are only able to determine the outcome at 72 hours, 30 days, and 1 year.
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
Participants
  Renal replacement therapy within 72 hours after liver transplant. | 8 | 13
  Renal replacement therapy at 30 days after liver transplant. | 8 | 5
  Renal replacement therapy at 1 year after liver transplant. | 7 | 9

7. Secondary Outcome: Persistent Renal Dysfunction
Description: Presence of a reduction in GFR by ≥ 25 mL/min or ≥ 50% from baseline at the time of follow-up. If patient died before the indicated follow-up time, the outcome was counted as positive (patient had persistent renal dysfunction).
Time Frame: 90 days and 1 year
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
Participants
  Persistent renal dysfunction at 90 days after liver transplant. | 24 | 25
  Persistent renal dysfunction at 1 year after liver transplant. | 28 | 32

8. Secondary Outcome: Serum Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: Change in serum NGAL levels from baseline to 2 hours after reperfusion of the portal vein (final - initial).
Time Frame: Baseline (start of surgery) and 2 hours after reperfusion of the portal vein
Population: Serum for NGAL determination was only collected at the coordinating center. It was not feasible to collect serum for all patients due to research personnel being unavailable during some off-hours and weekend liver transplants.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 37 | 38
ng/mL | 20.8 [1.8 to 61.4] | 26.15 [7.0 to 44.9]

9. Secondary Outcome: Urine Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: Change in urine NGAL levels from baseline to 2 hours after reperfusion of the portal vein (final - initial).
Time Frame: Baseline (start of surgery) and 2 hours after reperfusion of the portal vein
Population: Urine for NGAL determination was only collected at the coordinating center. It was not feasible to collect urine for all patients due to research personnel being unavailable during some off-hours and weekend liver transplants.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 39 | 40
ng/mL | 156.3 [8.2 to 491.7] | 81.85 [5.8 to 250.2]

10. Other Pre Specified Outcome: Blood Product Transfusions
Description: The number of units of packed red blood cells, fresh frozen plasma, platelets, and cryoprecipitate transfused during surgery. We had originally proposed to measure up until 72 hours after surgery, but we were not able to collect this data at all centers. Therefore, only blood product transfusions during surgery are reported.
Time Frame: During surgery
Population: Intention-to-treat population. Excludes participants that were withdrawn after randomization.
Measure: Median (Inter-Quartile Range); unit: Units of blood product transfused
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
Number analyzed (Participants) | 86 | 85
Units of blood product transfused
  Packed red blood cells | 4 [1 to 7] | 5 [1 to 8]
  Fresh frozen plasma | 8.5 [3 to 14] | 9 [3 to 18]
  Platelets | 2 [0 to 2] | 2 [0 to 3]
  Cryoprecipitate | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of enrollment until the end of liver transplantation surgery, with the exception of surgical site infection which was assessed until 2 weeks after surgery. Serious adverse events were assessed until 2 weeks after surgery. Deaths were assessed for up to 1 year (see Outcome Measures: Patient survival).
Description: Adverse events were defined as any untoward or unfavorable event that is outside that normally expected for the clinical course of liver transplantation, as reported by the study clinicians (attending anesthesiologist or surgeon) or the site prinicipal investigator.
Arm/Group | Mild Hypothermia & Esophageal Cooling/Warming Device | Normothermia & Esophageal Cooling/Warming Device
All-Cause Mortality (participants affected / at risk) | 5/86 | 7/85
Serious Adverse Events (participants affected / at risk) | 5/86 | 3/85
Other Adverse Events (participants affected / at risk) | 15/86 | 15/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hypothermia & Esophageal Cooling/Warming Device (N=86) | Normothermia & Esophageal Cooling/Warming Device (N=85)
Primary non-function of the liver (Hepatobiliary disorders) | 1 (1) | 1 (1) — Retransplantation within 7 days
Inferior vena cava thrombus (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intraoperative cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Disseminated fungal infection leading to death (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hypothermia & Esophageal Cooling/Warming Device (N=86) | Normothermia & Esophageal Cooling/Warming Device (N=85)
Bleeding (significant) with refractory severe coagulopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — Bleeding not attributable to vascular injury. Ongoing clinical coagulopathy, or lab evidence of persistent INR > 4 or fibrinogen < 75 mg/dL, despite aggressive treatment (15 mL/kg FFP, cryo 10 units x 2 doses, and antifibrinolytics).
Bleeding, upper gastrointestinal with esophageal temperature management device insertion (Gastrointestinal disorders) | 0 (0) | 0 (0) — Blood return > 500mL at time of esophageal temperature management device insertion
Hypothermia, severe (General disorders) | 1 (1) | 0 (0) — Temperature < 33 deg C for > 30 min
Oropharyngeal, dental, or esophageal trauma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Perforation or damage to esophageal temperature management device (Product Issues) | 0 (0) | 0 (0)
Cardiac arrhythmia (Cardiac disorders) | 2 (2) | 1 (1) — Intraoperative arrhythmia requiring treatment, excluding bradycardia at the time of liver reperfusion.
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Surgical bleeding, severe (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) — Not attributable to coagulopathy
Postreperfusion syndrome (Hepatobiliary disorders) | 1 (1) | 2 (2) — Subjective, as reported by attending anesthesiologist
Esophageal temperature management device problem (Product Issues) | 2 (2) | 1 (1) — Inadequate gastric suction or decompression, or accidental tracheal extubation during manipulation.
Electrolytes, overcorrection of hyponatremia (Renal and urinary disorders) | 0 (0) | 1 (1) — 1.5 mEq/L/h increase during surgery
Portal vein thrombus (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Drug error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cisatracurium concentration higher than expected (10 mg/mL instead of 2 mg/mL)
Traumatic central line insertion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Right internal jugular vein traumatic insertion and dilation
Cardiovascular event, non-serious (Cardiac disorders) | 1 (1) | 1 (1) — Self-limited unexplained hypotension or bradycardia, not requiring treatment.
Surgical site infection (Infections and infestations) | 0 (0) | 2 (2) — Within 2 weeks of surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT03534141/Prot_SAP_000.pdf